CLINICAL TRIAL: NCT02645604
Title: Artemether-Lumefantrine Resistance Monitoring in Children With Uncomplicated Plasmodium Falciparum Malaria in Mali
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999916033; 16-I-N033
Record Dates: First submitted 2016-01-01; First posted 2016-01-05 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2018-12-14

CONDITIONS: Accute Falciparum Malaria
Keywords: Artemisinin Combination Therapy (ACT)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
Background: Malaria is a disease caused by a parasite. People get malaria if they are bitten by an parasite-infected mosquito. A drug called artemether-lumefantrine (AL) can treat malaria. Although iAL has helped make the malaria problem less severe in the African country of Mali, researchers want to find out if malaria parasites are becoming resistant to this drug.

Objective: To test for AL-resistant parasites in children with malaria in Mali.

Eligibility:

AL resistance monitoring study: children aged 2 17 years who live in Kenieroba, Mali, and have malaria.

Blood collection substudy: healthy volunteers aged 18 65 years.

Design:

Volunteers for the substudy will have blood taken up to 6 times a year.

Study participants will be screened with 1 finger-prick blood sample. Girls may have a pregnancy test.

Baseline visit: Participants will have a physical exam. Their vital signs and temperature will be measured. They will answer questions about their symptoms. They will give a blood sample.

Participants will get 6 doses of AL over 3 days. They will take it in tablet form with milk.

Some participants will also stay at the clinic for 2 days. They will have a catheter placed in a vein. They will have blood taken frequently.

Participants will have follow-up visits for about 1 month. They may have:

Physical exam performed

Vital signs and temperature measured

Symptom questionnaire administered

Finger-prick blood sample and/or a regular blood sample taken

Pregnancy test given

Antimalarial medications other than AL provided.

DETAILED DESCRIPTION:
Artemether-lumefantrine (AL) has replaced artesunate + amodiaquine as the frontline artemisinin (ART) combination therapy (ACT) for uncomplicated Plasmodium falciparum malaria in Mali. It is not known whether parasites are developing resistance to AL in Mali, where we are studying how naturally-acquired immunity and sickle-cell trait reduce malaria risk and parasite density in our pediatric study population. AL Resistance Monitoring Study: To monitor for emerging AL resistance in vivo and lumefantrine (LF) resistance ex vivo, we will conduct a standard WHO-recommended protocol to measure AL resistance rates over the next 4 years. We will enroll all children aged 2-17 years with uncomplicated falciparum malaria and parasite count between 2,000 and 200,000 parasites per microliter, treat them with AL on D0, D1, and D2, confirm adequate LF plasma concentrations on Day 7, and monitor for malaria symptoms and recurrent parasitemias on D0, D1, D2, D3, D7, D14, D21, and D28. In related laboratory studies, we will use blood samples taken at the times of enrollment and recrudescence to measure parasite susceptibility to LF and other antimalarial drugs ex vivo; investigate genetic and transcriptional determinants of parasite response to AL in vivo and LF ex vivo; and prepare cryopreserved parasites for future work on drug action and resistance mechanisms. Parasite Clearance Substudy: We have recently discovered an agedependent acceleration of parasite clearance rates in Malian children, and postulate that it is mediated by IgG specific for Plasmodium falciparum erythrocyte membrane protein 1 (PfEMP1), the parasite s main virulence factor on the surface of infected red blood cells (iRBCs). We hypothesize that ART exposure induces the premature expression of PfEMP1 on the surface of circulating ring-iRBCs in vivo. To test this hypothesis, we will calculate parasite clearance rates in a subset of subjects with relatively high parasite densities, and relate these rates to the ability of autologous IgG to recognize ring-iRBCs over the first 8 hours of ART exposure in vivo. In this same subset of patients, we will also explore whether AL induces parasite dormancy in vivo by removing parasites at H0, H6, H24, H48, D3, D7, and D14 following AL therapy, and cloning them to quantify the number of viable parasites. Blood Collection Study: We have found that sickle-cell trait (HbAS), like naturally-acquired humoral immunity, reduces both malaria risk and parasite density in our study population, and that this protection is associated with abnormal PfEMP1 display on the iRBC surface. To elucidate the molecular mechanism of this phenotype and explore how it may synergize with naturally-acquired IgG responses, we will investigate whether the development of PfEMP1 trafficking machinery is impaired in HbAS compared to normal homozygous hemoglobin A (HbAA) red blood cells (RBCs). To test this, we will purify parasite isolates from children with malaria, inoculate them into HbAA and HbAS RBCs from healthy adult donors, and follow their intraerythrocytic development using flow cytometry and electron microscopy.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subject Inclusion Criteria: AL Resistance Monitoring Study

* Resident of Kenieroba
* Age 2 to 17 years
* Uncomplicated falciparum malaria, confirmed by the presence of asexual P. falciparum parasites on blood film
* Asexual P. falciparum count between 2,000 and 200,000/ microliters (inclusive) at screening
* Tympanic or axillary temperature greater than or equal to 37.5 (Infinite)C or history of fever in the previous 24 hours
* Written informed consent from the child s parent or guardian, and assent from children aged 14-17 years

Subject Inclusion Criteria: Parasite Clearance Substudy

* Enrolled in the AL Resistance Monitoring Study
* Asexual P. falciparum count greater than or equal to 10,000/ microliters at screening
* Hb level greater than or equal to 7 g/dL

Subject Inclusion Criteria: Blood Collection Study

* Age 18 to 65 years or 5 to 65 years old for the mosquito infectivity study
* Healthy-appearing
* Hb level greater than or equal to 7 g/dL

EXCLUSION CRITERIA:

Subject Exclusion Criteria: AL Efficacy Study

* Signs of severe malaria, defined as one or more of the following:

  * Blantyre Coma Scale less than or equal to 3/5 in children
  * Witnessed convulsions
  * Severe prostration
  * Shock (poor perfusion, cool peripheries)
  * Hb <5 g/dL
  * Jaundice
  * Respiratory distress (labored breathing, nasal flaring, intercostal retraction)
  * Anuria for 24 hours or more
  * Repetitive vomiting
  * Cessation of eating and drinking
* Acute illness other than uncomplicated falciparum malaria requiring treatment
* Presence of P. ovale or P. malariae parasites on blood film
* Severe malnutrition: http://www.who.int/childgrowth/standards/Technical_report.pdf
* Pregnancy or breastfeeding an infant
* Planning to become pregnant in the next 1 month
* History of taking an ACT in the previous 14 days
* Known hypersensitivity to artemether or LF
* Co-administration of strong inducers of CYP3A4 such as rifampin, carbamazepine, phenytoin, and St. John s wort
* Splenectomy
* Any condition that in the opinion of the investigator would render the patient unable to comply with the protocol (e.g., psychiatric disease)
* Any health condition that in the opinion of the investigator would confound data analysis (e.g., HIV infection) or pose unnecessary exposure risks to the subject

Subject Exclusion Criteria: Parasite Clearance Substudy

-Prior enrollment in the Parasite Clearance Substudy in current transmission season

Subject Exclusion Criteria: Blood Collection Study

* P. falciparum infection, as determined by thick blood smear examination (unless the subject is being screened for inclusion in the mosquito infectivity study, in which case parasitemia, as detected by RDT or smear, is an inclusion criteria)
* History of taking an ACT in the previous 28 days

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2016-01-01; Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Treatment failure up to Day 28. A subject will be defined as a treatment failure if the subject has developed P. falciparum parasitemia detected by thick blood smear (not by PCR) between the time that parasitemia becomes undetectable and Day 28,... | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Rick M Fairhurst, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Malaria Research and Training Center, Bamako, Mali

REFERENCES:
- [Background] Lopera-Mesa TM, Doumbia S, Chiang S, Zeituni AE, Konate DS, Doumbouya M, Keita AS, Stepniewska K, Traore K, Diakite SA, Ndiaye D, Sa JM, Anderson JM, Fay MP, Long CA, Diakite M, Fairhurst RM. Plasmodium falciparum clearance rates in response to artesunate in Malian children with malaria: effect of acquired immunity. J Infect Dis. 2013 Jun 1;207(11):1655-63. doi: 10.1093/infdis/jit082. Epub 2013 Feb 28. PMID 23448727
- [Background] Ndour PA, Lopera-Mesa TM, Diakite SA, Chiang S, Mouri O, Roussel C, Jaureguiberry S, Biligui S, Kendjo E, Claessens A, Ciceron L, Mazier D, Thellier M, Diakite M, Fairhurst RM, Buffet PA. Plasmodium falciparum clearance is rapid and pitting independent in immune Malian children treated with artesunate for malaria. J Infect Dis. 2015 Jan 15;211(2):290-7. doi: 10.1093/infdis/jiu427. Epub 2014 Sep 2. PMID 25183768
- [Background] Worldwide Antimalarial Resistance Network (WWARN) AL Dose Impact Study Group. The effect of dose on the antimalarial efficacy of artemether-lumefantrine: a systematic review and pooled analysis of individual patient data. Lancet Infect Dis. 2015 Jun;15(6):692-702. doi: 10.1016/S1473-3099(15)70024-1. Epub 2015 Mar 16. PMID 25788162
- [Derived] Petersen JEV, Saelens JW, Freedman E, Turner L, Lavstsen T, Fairhurst RM, Diakite M, Taylor SM. Sickle-trait hemoglobin reduces adhesion to both CD36 and EPCR by Plasmodium falciparum-infected erythrocytes. PLoS Pathog. 2021 Jun 11;17(6):e1009659. doi: 10.1371/journal.ppat.1009659. eCollection 2021 Jun. PMID 34115805